CLINICAL TRIAL: NCT05461651
Title: Prospective, Randomized, Double Blinded Trial Comparing Clinical, Radiological and Laboratory Outcomes in Prevention of Infection After Total Knee Arthroplasty With or Without Vancomycin.
Brief Title: Infection Prevention After TKA With or Without Vancomycin
Acronym: TKA_Vanco
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Principal Investigator, Rafał Kamiński, Professor, Centre of Postgraduate Medical Education
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TKA
Record Dates: First submitted 2022-02-03; First posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Infection
Keywords: TKA, Vancomycin
MeSH Terms: conditions — Infections | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Knee arthroplasty (Sham Comparator): Knee arthroplasty without addition of antibiotic wash oraz antibitiotic powder to the surgery site
  Interventions: Procedure: Knee arthroplasty
- Knee arthroplasty + vancomycin (Active Comparator): Knee arthroplasty with addition of vancomysin powder to the surgery site
  Interventions: Procedure: Knee arthroplasty

INTERVENTIONS:
Procedure: Knee arthroplasty — total or unilateral knee arthroplasty

SUMMARY:
Prospective, Randomized, Double Blinded Trial Comparing Clinical, Radiological and Laboratory Outcomes in prevention of infection after Total Knee Arthroplasty With or Without Vancomycin.

DETAILED DESCRIPTION:
Infection after surgery is one of the most common complication after total knee replacement. Our prospective randomized study is intended to show if addition of vancomycin to the joint before the wound closure will decrease infection after operation.

ELIGIBILITY:
Inclusion Criteria:

* Gosnartrosis

Exclusion Criteria:

* no informed consent to participate in the study age under 40 multilligament injury or single plane knee instability another musculoskeletal disorders in lower limb ASA score > II

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of surgical site infection | up to 24 months
  The incidence of deep and superficial SSI after knee arthroplasty

SECONDARY OUTCOMES:
Blood test - CRP | 12 weeks,
  inflammatory reaction - CRP
Blood test - IL 6 | 12 weeks,
  inflammatory reaction - Il-6
Functional tests | 12 weeks,
  hop-for-distance
Functional tests | 6 months,
  hop-for-distance
Functional tests | 12 months
  hop-for-distance
Functional tests | 24 months
  hop-for-distance
Knee injury and Osteoarthritis Outcome Score | 6 weeks
  Knee Injury and Osteoarthritis Outcome Score; KOOS is intended to be used for knee injury that can result in post traumatic osteoarthritis (OA); KOOS has high test-retest reliability. In patients with knee injury, ICCs for the Pain subscale range from 0.85-0.93, the Symptoms subscale from 0.83-0.95, the ADL subscale from 0.75-0.91, the Sport/Rec subscale from 0.61-0.89 and the QOL subscale from 0.83-0.95. In patients with knee OA, ICCs for the Pain subscale range from 0.8-0.97, the Symptoms subscale from 0.74-0.94, the ADL subscale from 0.84-0.94, the Sport/Rec subscale from 0.65-0.92 and the QOL subscale from 0.6-0.91 (4).
Knee injury and Osteoarthritis Outcome Score | 6 months
  Knee Injury and Osteoarthritis Outcome Score; KOOS is intended to be used for knee injury that can result in post traumatic osteoarthritis (OA); KOOS has high test-retest reliability. In patients with knee injury, ICCs for the Pain subscale range from 0.85-0.93, the Symptoms subscale from 0.83-0.95, the ADL subscale from 0.75-0.91, the Sport/Rec subscale from 0.61-0.89 and the QOL subscale from 0.83-0.95. In patients with knee OA, ICCs for the Pain subscale range from 0.8-0.97, the Symptoms subscale from 0.74-0.94, the ADL subscale from 0.84-0.94, the Sport/Rec subscale from 0.65-0.92 and the QOL subscale from 0.6-0.91 (4).
Knee injury and Osteoarthritis Outcome Score | 12 months
  Knee Injury and Osteoarthritis Outcome Score; KOOS is intended to be used for knee injury that can result in post traumatic osteoarthritis (OA); KOOS has high test-retest reliability. In patients with knee injury, ICCs for the Pain subscale range from 0.85-0.93, the Symptoms subscale from 0.83-0.95, the ADL subscale from 0.75-0.91, the Sport/Rec subscale from 0.61-0.89 and the QOL subscale from 0.83-0.95. In patients with knee OA, ICCs for the Pain subscale range from 0.8-0.97, the Symptoms subscale from 0.74-0.94, the ADL subscale from 0.84-0.94, the Sport/Rec subscale from 0.65-0.92 and the QOL subscale from 0.6-0.91 (4).
Knee injury and Osteoarthritis Outcome Score | 24 months
  Knee Injury and Osteoarthritis Outcome Score; KOOS is intended to be used for knee injury that can result in post traumatic osteoarthritis (OA); KOOS has high test-retest reliability. In patients with knee injury, ICCs for the Pain subscale range from 0.85-0.93, the Symptoms subscale from 0.83-0.95, the ADL subscale from 0.75-0.91, the Sport/Rec subscale from 0.61-0.89 and the QOL subscale from 0.83-0.95. In patients with knee OA, ICCs for the Pain subscale range from 0.8-0.97, the Symptoms subscale from 0.74-0.94, the ADL subscale from 0.84-0.94, the Sport/Rec subscale from 0.65-0.92 and the QOL subscale from 0.6-0.91 (4).
36-Item Short Form Survey | 6 weeks
  Quality of life, pain SF-36
36-Item Short Form Survey | 6 months
  Quality of life, pain SF-36
36-Item Short Form Survey | 12 months
  Quality of life, pain SF-36
36-Item Short Form Survey | 24 months
  Quality of life, pain SF-36
Visual analog Scale | 6 weeks
  Pain Visual Analog Scale
  The pain VAS is a unidimensional measure of pain intensity. The most simple VAS is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptom, pain, health)[8] orientated from the left (worst) to the right (best).
Visual analog Scale | 6 months
  Pain Visual Analog Scale
  The pain VAS is a unidimensional measure of pain intensity. The most simple VAS is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptom, pain, health)[8] orientated from the left (worst) to the right (best).
Visual analog Scale | 12 months
  Pain Visual Analog Scale
  The pain VAS is a unidimensional measure of pain intensity. The most simple VAS is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptom, pain, health)[8] orientated from the left (worst) to the right (best).
Visual analog Scale | 24 months
  Pain Visual Analog Scale
  The pain VAS is a unidimensional measure of pain intensity. The most simple VAS is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptom, pain, health)[8] orientated from the left (worst) to the right (best).
Tegner Lysholm Knee Scoring Scale | 6 weeks
  The Lysholm Knee Scoring Scale is a patient-reported instrument that consists of subscales for pain, instability, locking, swelling, limp, stair climbing, squatting, and the need for support. Scores range from 0 (worse disability) to 100 (less disability).
Tegner Lysholm Knee Scoring Scale | 6 months
  The Lysholm Knee Scoring Scale is a patient-reported instrument that consists of subscales for pain, instability, locking, swelling, limp, stair climbing, squatting, and the need for support. Scores range from 0 (worse disability) to 100 (less disability).
Tegner Lysholm Knee Scoring Scale | 12 months
  The Lysholm Knee Scoring Scale is a patient-reported instrument that consists of subscales for pain, instability, locking, swelling, limp, stair climbing, squatting, and the need for support. Scores range from 0 (worse disability) to 100 (less disability).
Tegner Lysholm Knee Scoring Scale | 24 months
  The Lysholm Knee Scoring Scale is a patient-reported instrument that consists of subscales for pain, instability, locking, swelling, limp, stair climbing, squatting, and the need for support. Scores range from 0 (worse disability) to 100 (less disability).

CONTACTS AND LOCATIONS:
Overall Officials: Rafal KAminski, Study Chair — CMKP
Locations (1):
- Department of Orthopaedics and Traumatology, Postgraduate Center for Medical Education, Professor A. Gruca Teaching Hospital, Otwock, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No